CLINICAL TRIAL: NCT01675557
Title: Pharmacokinetic Comparison of Vitamin's D2 and D3 in Stage 5 Chronic Kidney
Brief Title: Pharmacokinetic Comparison of Vitamin's D2 and D3 in Stage 5 Chronic Kidney Disease Patients on Chronic Hemodialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Creighton15
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Chronic Kidney Disease
Keywords: chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Cholecalciferol; Ergocalciferols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vitamin D2 (Active Comparator): a single oral dose of vitamin D2
  Interventions: Dietary Supplement: Vitamin D2
- Placebo (Placebo Comparator): a single oral dose of a placebo
  Interventions: Dietary Supplement: Placebo
- Vitamin D3 (Experimental): A single oral dose of vitamin D3
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — a single oral dose of vitamin D3
  Other Names: Cholecalciferol
  Arms: Vitamin D3
Dietary Supplement: Vitamin D2 — a single oral dose of vitamin D2
  Other Names: ergocalciferol
  Arms: Vitamin D2
Dietary Supplement: Placebo — a single oral dose of placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the pharmacokinetic 25(OH)D and 1,25(OH)2D responses to a single oral dose of vitamin D2 or vitamin D3 in a group of Stage 5-Chronic Kidney Disease subjects requiring chronic hemodialysis.

DETAILED DESCRIPTION:
This is a randomized, single blind, controlled study. Subjects will be randomly assigned to receive 1) placebo capsules (control group); 2) capsules with ergocalciferol (the vitamin D2 group); or 3) capsules with cholecalciferol (the vitamin D3 group).

ELIGIBILITY:
Inclusion Criteria:

* 30 men and women, ages 20-65, BMI 18-30, requiring chronic hemodialysis

Exclusion Criteria:

* They will habitually consume less than 16 oz of milk per day and get less than 10 hours of sun exposure per week. We will exclude those with granulomatous conditions, cirrhotic liver disease, and those taking anticonvulsants, barbiturates, or steroids in any form or any investigational drugs within 4 weeks. We will exclude those with pregnancy or planned pregnancy, hypercalcemia (>10.4 mg/dl) previously recorded, chronic GI disease which would interfere with absorption, any allergy to vitamin D3, or chronic vitamin D intake >1,000 IU daily. Subjects will continue to take a calcitriol analogue and phosphorus binder as prescribed by their nephrologist. Calcitriol analogues are to be documented and remain constant throughout study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
25(OH)D | 16 weeks
  25(OH)D levels will be drawn at intervals over 16 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Laura AG Armas, MD,MS, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Graeff-Armas LA, Kaufmann M, Lyden E, Jones G. Serum 24,25-dihydroxyvitamin D3 response to native vitamin D2 and D3 Supplementation in patients with chronic kidney disease on hemodialysis. Clin Nutr. 2018 Jun;37(3):1041-1045. doi: 10.1016/j.clnu.2017.04.020. Epub 2017 Apr 30. PMID 28506446